CLINICAL TRIAL: NCT00145574
Title: Randomized, Double-blind, Placebo-controlled Efficacy and Safety Study of Colesevelam HCl Administered to Pediatric Patients With Heterozygous Familial Hypercholesterolemia on a Stable Dose of Statins or Treatment Naive to Lipid-lowering Therapy
Brief Title: Efficacy and Safety of Colesevelam in Pediatric Patients With Genetic High Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Michael Melino, Daiichi Sankyo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-410
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Hypercholesterolemia
Keywords: Pediatric; hypercholesterolemia; colesevelam
MeSH Terms: conditions — Hypercholesterolemia | interventions — Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- high dose colesevelam (Experimental): colesevelam HCl 3.750 g
  Interventions: Drug: colesevelam HCl
- Low dose colesevelam (Experimental): Low dose colesevelam 1.875 g
  Interventions: Drug: colesevelam HCl
- placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: colesevelam HCl — Tablets
  Arms: Low dose colesevelam; high dose colesevelam
Drug: placebo — Matching Tablets
  Arms: placebo

SUMMARY:
This study will evaluate the lipid-lowering effect and safety of colesevelam therapy administered to heterozygous familial pediatric patients 10 through 17 years of age who are on a stable dose of a pediatric-approved statin monotherapy (atorvastatin, lovastatin, simvastatin or pravastatin), or who are treatment naive to lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Ages 10 to 17 years inclusive
* Diagnosis of heterozygous familial hypercholesterolemia
* On a stable dose of statin monotherapy or are treatment naive to lipid- lowering agents
* On a low-cholesterol diet

Exclusion Criteria:

* Patients should not have serious concomitant conditions that could interfere with the analysis of the results or that could interfere with the well-being of the patients

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (8):
  - Washington D.C., District of Columbia
  - St Louis, Missouri
  - New Hyde Park, New York
  - New York, New York
  - The Bronx, New York
  - Cincinnati, Ohio
  - Wexford, Pennsylvania
  - Salt Lake City, Utah
- Camperdown NSW, Australia
- Vienna, Austria
- Canada (5):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Laval, Quebec
  - Stefoy, Quebec
- Israel (4):
  - Holon
  - Jerusalem
  - Kefer Saba
  - Tel Litwinsky
- Netherlands (2):
  - Amsterdam
  - Rotterdam
- Oslo, Norway
- South Africa (3):
  - Observatory
  - Pretoria
  - Tygerberg

REFERENCES:
- [Derived] Stein EA, Marais AD, Szamosi T, Raal FJ, Schurr D, Urbina EM, Hopkins PN, Karki S, Xu J, Misir S, Melino M. Colesevelam hydrochloride: efficacy and safety in pediatric subjects with heterozygous familial hypercholesterolemia. J Pediatr. 2010 Feb;156(2):231-6.e1-3. doi: 10.1016/j.jpeds.2009.08.037. Epub 2009 Oct 31. PMID 19879596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 41 clinical sites; Australia (1 site), Austria (1 site), Canada (5 sites), Hungary (1 site), Israel (5 sites), New Zealand (1 site), Norway (2 sites), Slovakia (3 sites), South Africa (4 sites), Czech Republic (3 sites), Netherlands (2 sites), and USA (13 sites). Study initiated November 5, 2005 completed December 18, 2007.
Pre-assignment Details: Period I Run-In (4 weeks): Period I was a single-blind stabilization period prior to randomization. All subjects received 6 placebo tablets daily. Objective was to evaluate dosing compliance and tolerability to the tablets prior to randomization. Subjects could be on stable pediatric approved statin regimen and low cholesterol diet for 6 weeks.
Groups:
- Placebo: Placebo similar to active
- Low Dose Colesevelam: Low dose colesevelam 1.9 grams per day
- High Dose Colesevelam: High dose colesevelam 3.8 grams per day
Period: Double Blind
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Started | 65 | 65 | 64
Completed | 64 | 60 | 62
Not Completed | 1 | 5 | 2
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — required restricted medicine | 0 | 1 | 0
Period: Open Label Long-term Extension
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Started | 0 | 0 | 184 (2 participants discontinued after completing double-blind but before starting open label.)
Completed | 0 | 0 | 173
Not Completed | 0 | 0 | 11
Not completed — Adverse Event | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — required restricted medicine | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | Total
Number analyzed (Participants) | 65 | 65 | 64 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 65 | 65 | 64 | 194
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.74) | 14.1 (2.19) | 13.9 (2.0) | 14.1 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 24 | 71
  Male | 44 | 39 | 40 | 123
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 15 | 45
  Canada | 7 | 9 | 7 | 23
  Austria | 0 | 1 | 0 | 1
  South Africa | 18 | 16 | 17 | 51
  Israel | 6 | 6 | 4 | 16
  Norway | 3 | 3 | 4 | 10
  Netherlands | 3 | 3 | 4 | 10
  Hungary | 6 | 7 | 6 | 19
  New Zealand | 2 | 1 | 2 | 5
  Slovakia | 2 | 0 | 2 | 4
  Czech Republic | 2 | 5 | 3 | 10
Statin Status [Number; unit: participants] — Non-naive refers to the number of participants who are taking statins. Naive refers to the number of participants who are not taking statins.
  participants
    non-naive | 48 | 50 | 49 | 147
    naive | 17 | 15 | 15 | 47
Tanner Stage [Number; unit: participants] — Tanner Stage represents a scale measuring physical development in children based on primary and secondary sexual characteristics. The scale has five stages, with Stage I representing prepuberty and Stage 5 representing adult physical development. Please refer to Tanner, JM; Growth at Adolescence, @nd ed. Oxford, England, Blackwell Scientific Publications, 1962 for complete definitions of each Tanner Stage of development.
  participants
    I | 0 | 0 | 0 | 0
    II | 9 | 15 | 15 | 39
    III | 20 | 16 | 16 | 52
    IV | 23 | 19 | 20 | 62
    V | 13 | 15 | 13 | 41
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index (BMI) kg/m2
  kg/m2 | 21.9 (4.30) | 23.4 (6.14) | 22.2 (4.75) | 22.5 (5.14)
height [Mean (Standard Deviation); unit: cm] — height in centimeters (cm)
  cm | 164.8 (10.35) | 160.7 (10.90) | 162.1 (11.94) | 162.5 (11.16)
weight [Mean (Standard Deviation); unit: kg] — mean weight in kilograms (kg) and standard deviation (SD)
  kg | 60.3 (15.32) | 61.5 (20.77) | 59.0 (16.81) | 60.3 (17.72)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Plasma Low Density Lipoprotein-cholesterol (LDL-C) From Day 1 (Study Baseline) to Week 8.
Description: Percent change in LDL-C (mg/dL) and standard deviation (SD) from Day 1 (Study Baseline)to Week 8 (last observation carried forward - LOCF)- Intent-to-Treat ITT population.
Time Frame: 8 weeks (week 8 - day 1)
Population: Intent-to-Treat Population for Double blind Period. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Number analyzed (Participants) | 65 | 63 | 63
percent change from baseline | 2.9 (16.46) | -3.7 (18.36) | -10.6 (19.36)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Colesevelam; The primary null hypotheses were tested sequentially in the following order: 1) no difference between the high-dose colesevelam HCl and placebo for percent change in LDL-C from study baseline to Week 8 endpoint with the last observation carried forward (LOCF) and 2) no difference between the low-dose colesevelam HCl and placebo for percent change in LDL-C from study baseline to Week 8 endpoint with LOCF. The hypotheses were tested at a 2-sided significance level of 5%; Test type: Superiority or Other; p = 0.1122, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs High Dose Colesevelam; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Percent Change in Plasma Total Cholesterol (TC) From Day 1 (Study Baseline) to Week 8.
Description: Percent change in total cholesterol (mg/dL) and standard deviation (SD) from Day 1 (Study Baseline) to Week 8 (last observation carried forward - LOCF)- Intent-to-Treat ITT population.
Time Frame: 8 weeks (week 8 - day 1)
Population: Intent-to-Treat Population for Double blind Period. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Number analyzed (Participants) | 65 | 63 | 63
percent change from baseline | 2.9 (13.29) | -1.1 (14.22) | -5.4 (15.8)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Colesevelam; Test type: Superiority or Other; p = 0.5260, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs High Dose Colesevelam; Test type: Superiority or Other; p = 0.0085, ANCOVA

3. Secondary Outcome: Percent Change in Plasma Triglycerides (TG) From Day 1 (Study Baseline) to Week 8.
Description: Percent change in triglycerides (mg/dL) and standard deviation (SD) from Day 1 (Study Baseline) to Week 8 (last observation carried forward - LOCF)- Intent-to-Treat ITT population.
Time Frame: 8 weeks (week 8 - day 1)
Population: Intent-to-Treat Population for Double blind Period. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Number analyzed (Participants) | 65 | 63 | 63
percent change from baseline | 12.5 (40.8) | 16.9 (35.7) | 12.5 (53.2)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Colesevelam; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs High Dose Colesevelam; Test type: Superiority or Other; p = 0.0008, ANCOVA

4. Secondary Outcome: Percent Change in Plasma High-density Lipoprotein-cholesterol (HDL-C) From Day 1 (Study Baseline) to Week 8.
Description: Percent change in HDL-C (mg/dL) and standard deviation (SD) from Day 1 (Study Baseline) to Week 8 (last observation carried forward - LOCF)- Intent-to-Treat ITT population.
Time Frame: 8 weeks (week 8 - day 1)
Population: Intent-to-Treat Population for Double blind Period. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Number analyzed (Participants) | 65 | 63 | 63
percent change from baseline | 2.5 (12.52) | 3.9 (12.45) | 8.5 (14.72)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Colesevelam; Test type: Superiority or Other; p = 0.0155, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs High Dose Colesevelam; Test type: Superiority or Other; p < 0.0001, ANCOVA

5. Secondary Outcome: Percent Change in Plasma Non-high Density Lipoprotein-cholesterol (Non-HDL-C) From Day 1 (Study Baseline) to Week 8.
Description: Percent change in non-HDL-C (mg/dL) and standard deviation (SD) from Day 1 (Study Baseline) to Week 8 (last observation carried forward - LOCF)- Intent-to-Treat ITT population.
Time Frame: 8 weeks (week 8 - day 1)
Population: Intent-to-Treat Population for Double blind Period. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Number analyzed (Participants) | 65 | 63 | 63
percent change from baseline | 3.4 (16.01) | -2.1 (17.32) | -8.4 (18.28)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Colesevelam; Test type: Superiority or Other; p = 0.3482, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs High Dose Colesevelam; Test type: Superiority or Other; p = 0.0006, ANCOVA

6. Secondary Outcome: Percent Change in Plasma Apolipoprotien A-I (Apo A-1) From Day 1 (Study Baseline) to Week 8.
Description: Percent change in Apolipoprotien A-I (Apo A-1) (mg/dL) and standard deviation (SD) from Day 1 (Study Baseline) to Week 8 (last observation carried forward - LOCF)- Intent-to-Treat ITT population.
Time Frame: 8 weeks (week 8 - day 1)
Population: Intent-to-Treat (ITT) Population in Double blind Period. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Number analyzed (Participants) | 63 | 62 | 61
percent change from baseline | 4.4 (14.62) | 7.0 (13.96) | 11.2 (16.79)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Colesevelam; Test type: Superiority or Other; p = 0.0002, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs High Dose Colesevelam; Test type: Superiority or Other; p < 0.0001, ANCOVA

7. Secondary Outcome: Percent Change in Plasma Apolipoprotein B (Apo B) From Day 1 (Study Baseline) to Week 8.
Description: Percent change in Apo B (mg/dL) and standard deviation (SD) from Day 1 (Study Baseline) to Week 8 (last observation carried forward - LOCF)- Intent-to-Treat ITT population.
Time Frame: 8 weeks (week 8 - day 1)
Population: Intent-to-Treat (ITT) Population in Double blind Period. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam
Number analyzed (Participants) | 63 | 62 | 61
percent change from baseline | 2.3 (14.78) | -0.7 (16.52) | -7.0 (14.45)
Statistical Analysis 1: Comparison: Placebo vs Low Dose Colesevelam; Test type: Superiority or Other; p = 0.7433, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs High Dose Colesevelam; Test type: Superiority or Other; p = 0.0003, ANCOVA

8. Secondary Outcome: Percent Change in Low-density Lipoprotein Cholesterol (LDL-C) From Study Baseline (Day 1) to Week 26.
Description: Percent change in low-density lipoprotein cholesterol from baseline to Week 26 was calculated for subpopulations representing each assigned treatment group during the Double blind Period, and for the overall population in the Open Label Extension Period.
Time Frame: 26 weeks (week 26 - day 1)
Population: Intent-to-Treat (ITT) Population. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Placebo: A subpopulation of the All High Dose treatment regimen of the Open Label Extension period of participants who were randomized to placebo treatment during the Double blind Period.
- Low Dose Colesevelam: A subpopulation of the All High Dose treatment regimen of the Open Label Extension period of participants who were randomized to low dose colesevelam 1.9 grams per day treatment during the Double blind Period.
- High Dose Colesevelam: A subpopulation of the All High Dose treatment regimen of the Open Label Extension period of participants who were randomized to high dose colesevelam 3.8 grams per day treatment during the Double blind Period.
- All High Dose Colesevelam in Open Label Extension: Open Label Extension was an 18 week open-label treatment period. All participants were treated with 3750 mg colesevelam (high-dose).
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | All High Dose Colesevelam in Open Label Extension
Number analyzed (Participants) | 62 | 56 | 60 | 178
percent change from baseline | -11.9 (22.39) | -16.8 (19.85) | -13.5 (21.58) | -14.0 (21.32)

9. Secondary Outcome: Percent Change in Total Cholesterol From Study Baseline (Day 1) to Week 26.
Description: Percent change in total cholesterol (TC) from baseline to Week 26 was calculated for subpopulations representing each assigned treatment group during the Double blind Period, and for the overall population in the Open Label Extension Period.
Time Frame: 26 weeks (week 26 - day 1)
Population: Intent to treat population. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | All High Dose Colesevelam in Open Label Extension
Number analyzed (Participants) | 62 | 56 | 60 | 178
percent change from baseline | -7.5 (17.21) | -9.1 (16.91) | -7.5 (17.55) | -8.0 (17.15)

10. Secondary Outcome: Percent Change in Triglycerides From Study Baseline (Day 1) to Week 26.
Description: Percent change in triglycerides from baseline to Week 26 was calculated for subpopulations representing each assigned treatment group during the Double blind Period, and for the overall population in the Open Label Extension Period.
Time Frame: 26 weeks (week 26 - day 1)
Population: Intent to treat population. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | All High Dose Colesevelam in Open Label Extension
Number analyzed (Participants) | 62 | 56 | 60 | 178
percent change from baseline | -5.3 (59.1) | 19.5 (58.0) | 14.2 (64.5) | 11.5 (61.8)

11. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) From Study Baseline (Day 1) to Week 26.
Description: Percent change in high-density lipoprotein cholesterol from baseline to Week 26 was calculated for subpopulations representing each assigned treatment group during the Double blind Period, and for the overall population in the Open Label Extension Period.
Time Frame: 26 weeks (week 26 - day 1)
Population: Intent to treat population. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | All High Dose Colesevelam in Open Label Extension
Number analyzed (Participants) | 62 | 56 | 60 | 178
percent change from baseline | 6.6 (13.64) | 8.5 (20.33) | 9.3 (19.37) | 8.1 (17.86)

12. Secondary Outcome: Percent Change in Non-high-density Lipoprotein Cholesterol From Study Baseline (Day 1) to Week 26.
Description: Percent change in non-high-density lipoprotein cholesterol from baseline to Week 26 was calculated for subpopulations representing each assigned treatment group during the Double blind Period, and for the overall population in the Open Label Extension Period.
Time Frame: 26 weeks (week 26 - day 1)
Population: Intent to treat population. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | All High Dose Colesevelam in Open Label Extension
Number analyzed (Participants) | 61 | 56 | 60 | 177
percent change from baseline | -10.0 (21.04) | -13.2 (19.9) | -11.0 (20.80) | -11.3 (20.53)

13. Secondary Outcome: Percent Change in Apolipoprotein A-I From Study Baseline (Day 1) to Week 26.
Description: Percent change in apolipoprotein A-I from baseline to Week 26 was calculated for subpopulations representing each assigned treatment group during the Double blind Period, and for the overall population in the Open Label Extension Period.
Time Frame: 26 weeks (week 26 - day 1)
Population: Intent to treat population. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | All High Dose Colesevelam in Open Label Extension
Number analyzed (Participants) | 52 | 52 | 57 | 161
percent change from baseline | 4.7 (12.95) | 4.9 (14.86) | 7.2 (15.34) | 5.6 (14.40)

14. Secondary Outcome: Percent Change in Apolipoprotein B From Study Baseline (Day 1) to Week 26.
Description: Percent change in apolipoprotein B from baseline to Week 26 was calculated for subpopulations representing each assigned treatment group during the Double blind Period, and for the overall population in the Open Label Extension Period.
Time Frame: 26 weeks (week 26 - day 1)
Population: Intent to treat population. Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | Low Dose Colesevelam | High Dose Colesevelam | All High Dose Colesevelam in Open Label Extension
Number analyzed (Participants) | 52 | 52 | 57 | 161
percent change from baseline | -11.4 (16.86) | -11.3 (18.71) | -11.2 (17.86) | -11.3 (17.72)

ADVERSE EVENTS:
Groups:
- Placebo Double Blind Period: Placebo taken from day 1 to week 8.
- Low Dose Colesevelam Double Blind Period: Low dose colesevelam 1.9 grams per day taken from day 1 to week 8.
- High Dose Colesevelam Double Blind Period: High dose colesevelam 3.8 grams per day taken from day 1 to week 8.
- High Dose Colesevelam Open Label Extension: All participants of the Open Label Extension (weeks 8-26) took colesevelam 3.8 grams per day.
Arm/Group | Placebo Double Blind Period | Low Dose Colesevelam Double Blind Period | High Dose Colesevelam Double Blind Period | High Dose Colesevelam Open Label Extension
Serious Adverse Events (participants affected / at risk) | 3/65 | 3/65 | 0/64 | 0/184
Other Adverse Events (participants affected / at risk) | 20/65 | 25/65 | 14/64 | 71/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double Blind Period (N=65) | Low Dose Colesevelam Double Blind Period (N=65) | High Dose Colesevelam Double Blind Period (N=64) | High Dose Colesevelam Open Label Extension (N=184)
contusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
renal hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
poisoning deliberate (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nasopharyngeal cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Double Blind Period (N=65) | Low Dose Colesevelam Double Blind Period (N=65) | High Dose Colesevelam Double Blind Period (N=64) | High Dose Colesevelam Open Label Extension (N=184)
nasopharyngitis (Infections and infestations) | 3 | 4 | 4 | 10
upper respiratory infections NOS (Infections and infestations) | 3 | 1 | 1 | 9
ear infection NOS (Infections and infestations) | 3 | 1 | 0 | 3
gastrointestinal viral NOS (Infections and infestations) | 2 | 0 | 0 | 4
influenza (Infections and infestations) | 0 | 0 | 2 | 7
vomiting NOS (Gastrointestinal disorders) | 1 | 2 | 1 | 0
diarrhea NOS (Gastrointestinal disorders) | 2 | 0 | 1 | 2
nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 7
rhinitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 6
headache (Nervous system disorders) | 2 | 3 | 2 | 14
dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
fatigue (General disorders) | 1 | 3 | 2 | 0
blood creatine phosphokinase increased (Investigations) | 0 | 2 | 1 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
abdominal pain NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reflects the following restrictive language in the Clinical Study Agreements: "If identified by Daiichi Sankyo,Inc. (DSI), any of DSI's confidential information as defined herein shall be deleted…Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publication prepared by the Study Site."